CLINICAL TRIAL: NCT06289504
Title: An Open-label, One-sequence Cross-over, Single-centre Trial, Investigating the Influence of CagriSema on Pharmacokinetics and Pharmacodynamics of Warfarin and Pharmacokinetics of Atorvastatin in Participants With Overweight or Obesity
Brief Title: A Study on How CagriSema Affects Levels of Atorvastatin and Warfarin in the Blood of Participants With Excess Body Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-4694; U1111-1295-4056 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide; Atorvastatin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CagriSema +Atorvastatin + Warfarin (Experimental): Participants will receive a single dose of atorvastatin and a single dose of warfarin followed by a 16-week CagriSema dose escalation period and a 7-week CagriSema maintenance period. Participants will also receive a single dose of atorvastatin and a single dose of warfarin in the maintenance period.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide; Drug: Atorvastatin; Drug: Warfarin

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously once weekly.
Drug: Semaglutide — Semaglutide will be administered subcutaneously once weekly.
Drug: Atorvastatin — Atorvastatin will be administered as a single dose orally 2 times during the study.
Drug: Warfarin — Warfarin will be administered as a single dose orally 2 times during the study.

SUMMARY:
This study will look at how CagriSema affects the blood levels of atorvastatin and warfarin. The study will look at the levels of warfarin and atorvastatin in the blood before the participant starts taking CagriSema and if this changes after the participant has taken CagriSema. The study will also investigate the effect of warfarin before and after the participant takes CagriSema and assess if the injection site affects the level of CagriSema in the blood. The study will last for about 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Aged 18-65 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) between 27.0 and 39.9 kilograms per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Previous dosing in a study with an amylin analogue.
* Presence or history of pathological bleeding tendencies, recent serious bleeding, recent myopathy or rhabdomyolysis, malignant hypertension and any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions including type 1 or type 2 diabetes mellitus.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, or as judged by the investigator.
* Glycated haemoglobin (HbA1c) greater than or equal to (≥) 6.5 % (48 millimoles per mole [mmol/mol]) at screening.
* Activated partial thromboplastin time (APTT) less than (<) 22.1 seconds (lower normal limit [LNL]-0%) or APTT greater than (>) 28.1 seconds (upper limit of normal [UNL) +0%) at screening.
* Prothrombin time < 70% (LNL-0%) or prothrombin time > 130% (UNL-0%) at screening.
* Use of prescription medicinal products or non-prescription drugs, including any herbal medicine known to interfere with the metabolic cytochrome P450 (CYP) pathways, such as perikon (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae within 14 days (or within 5 half-lives of the medicinal product, whichever is longest) of screening, with the exception of use of routine vitamins (vitamins used within a normal dose reference interval), occasional use of paracetamol and highly effective contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
AUC0-72hours,atorv,SD: Area under the atorvastatin plasma concentration-time curve from time 0 to 72 hours after a single dose of atorvastatin without CagriSema exposure and at CagriSema steady state | Day 1 (pre-dose to 72 hours post-dose) and day 171 (pre-dose to 72 hours post-dose)
  Measured in hours*nanomoles per liter (hours*nmol/L).
AUC0-168hours,S-war,SD: Area under the S-warfarin plasma concentration-time curve from time 0 to 168 hours after a single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.

SECONDARY OUTCOMES:
AUC0-∞,atorv,SD: Area under the atorvastatin plasma concentration curve from time 0 to infinity after single dose of atorvastatin without CagriSema exposure and at CagriSema steady state | Day 1 (pre-dose to 72 hours post-dose) and day 171 (pre-dose to 72 hours post-dose)
  Measured in hours*nmol/L.
Cmax,atorv,SD: Maximum observed atorvastatin plasma concentration after single dose of atorvastatin without CagriSema exposure and at CagriSema steady state | Day 1 (pre-dose to 72 hours post-dose) and day 171 (pre-dose to 72 hours post-dose)
  Measured in nanomoles per liter (nmol/L).
tmax,atorv,SD: Time to maximum observed atorvastatin plasma concentration after single dose of atorvastatin without CagriSema exposure and at CagriSema steady state | Day 1 (pre-dose to 72 hours post-dose) and day 171 (pre-dose to 72 hours post-dose)
  Measured in hours.
AUC0-∞,S-war,SD: Area under the S-warfarin plasma concentration curve from time 0 to infinity after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
Cmax,S-war,SD: Maximum observed S-warfarin plasma concentration after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in nmol/L.
tmax,S-war,SD: Time to maximum observed S-warfarin plasma concentration after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in hours.
iAUCINR,0-168hours: Incremental area under the INR-curve from 0 to 168 hours after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
INRmax: Maximum observed INR response after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in ratio.
tINRmax: Time to maximum observed INR response after single dose of warfarin without CagriSema exposure and at CagriSema steady state | Day 8 (pre-dose to 168 hours post-dose) and day 178 (pre-dose to 168 hours post-dose)
  Measured in hours.
Rac,0-168hours,cagri: The ratio of the area under the cagrilintide plasma concentration curve from 0 to 168 hours after the 4th dose of CagriSema to the area under the plasma concentration curve from 0 to 168 hours after the 1st dose | Day 23 (pre-dose to 168 hours post-dose) and day 44 (pre-dose to 168 hours post-dose)
  Measured in ratio.
Rac,0-168hours,sema: The ratio of the area under the semaglutide plasma concentration curve from 0 to 168 hours after the 4th dose of CagriSema to the area under the plasma concentration curve from 0 to 168 hours after the 1st dose | Day 23 (pre-dose to 168 hours post-dose) and day 44 (pre-dose to 168 hours post-dose
  Measured in ratio.
AUC0-168hours, 4th dose cagri: Area under the cagrilintide plasma concentration curve from 0 to 168 hours after 4th dose of CagriSema | Day 44 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
AUC0-168hours,4th dose Sema: Area under the semaglutide plasma concentration curve from 0 to 168 hours after 4th dose of CagriSema | Day 44 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
AUC0-168hours, cagri 2.4mg, SS: Area under the cagrilintide plasma concentration curve from 0 to 168 hours at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
AUC0-168hours, sema 2.4mg, SS: Area under the semaglutide plasma concentration curve from 0 to 168 hours at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in hours*nmol/L.
Cmax, cagri, SS: Maximum observed cagrilintide plasma concentration at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in nmol/L.
tmax, cagri, SS: Time to maximum observed cagrilintide plasma concentration at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in hours.
Cmax, sema,SS: Maximum observed semaglutide plasma concentration at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in nmol/L.
tmax, sema, SS: Time to maximum observed semaglutide plasma concentration at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in hours.
CL/Fcagri,SS: total apparent clearance of cagrilintide at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in litres per hour (L/h).
CL/Fsema,SS: total apparent clearance of semaglutide at steady state | Day 163 (pre-dose to 168 hours post-dose)
  Measured in litres per hour (L/h).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com